CLINICAL TRIAL: NCT05849051
Title: Little Cigar and Cigarillo Warnings to Reduce Tobacco-Related Cancers and Disease: Randomized Controlled Trial Among US Adults Who Use LCCs
Brief Title: Little Cigar and Cigarillo Warnings Among US Adults Who Use LCCs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 22-2531; R01CA240732 (NIH)
Record Dates: First submitted 2023-04-26; First posted 2023-05-08 (Actual); Results first posted 2025-01-08 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: Tobacco Use
Keywords: Cigar Warnings; Little Cigar Use; Cigar Use; Cigarillo Use
MeSH Terms: conditions — Tobacco Use

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Newly developed warnings with images (Experimental): Participants receive newly developed warnings intervention
  Interventions: Behavioral: Newly developed warnings with images at 30% size
- FDA proposed text-only warnings (Experimental): Participants receive FDA proposed text only warning intervention
  Interventions: Behavioral: FDA proposed text-only warnings at 30% size
- Control group, no intervention (No Intervention): Participants do not receive an intervention

INTERVENTIONS:
Behavioral: Newly developed warnings with images at 30% size — On study days 1-6, 8-13 and 15-20, participants in this condition will view an image of a little cigar and cigarillo package with a warning developed by the study team that includes an image. The warnings will take up 30% of the package. Participants will view a total of 6 different warnings over the course of 6 days each week, this will be repeated 3 times during the study, resulting in a total of 18 exposures. Participants will be required to view the warning for at least 5 seconds.
  Arms: Newly developed warnings with images
Behavioral: FDA proposed text-only warnings at 30% size — On study days 1-6, 8-13 and 15-20, participants in this condition will view an image of a little cigar and cigarillo package with a warning proposed by the FDA which is text only. The warnings will take up 30% of the package. Participants will view a total of 6 different warnings over the course of 6 days each week, this will be repeated 3 times during the study, resulting in a total of 18 exposures. Participants will be required to view the warning for at least 5 seconds.
  Arms: FDA proposed text-only warnings

SUMMARY:
The goal of this research is to assess whether little Cigars and cigarillos (LCC) warnings developed by the study team are more effective than the current warnings proposed by FDA for LCC products. A 3-week web-based randomized controlled trial will be conducted in the United States. Participants are adult persons who currently use LCCs.

DETAILED DESCRIPTION:
In this study, LCC warnings on packs will be electronically presented to participants over time to determine if newly developed LCC warnings increase quit intentions compared to FDA-proposed text-only warnings and a control condition (in which participants do not see LCC packs or warnings.) A daily diary methodology will be employed to present LCC warnings on packs to participants over time. Qualtrics will contact, screen, consent, and administer the survey. To enroll participants, Qualtrics will screen participants using the inclusion criteria and measures and invite eligible participants to enroll in the study.

At the beginning of the baseline survey (day 0), participants will first consent to participate in the study and then complete a questionnaire about their tobacco use and behaviors (e.g., intentions and quit attempts) and other measures of interest. At the end of the baseline questionnaire, survey software will randomly assign participants to one of the 3 study conditions. The three study conditions are 1) Newly developed warnings with images (the six most effective warnings developed by the study team), 2) FDA-proposed text-only warnings, or 3) control condition in which participants will not receive an intervention (no warnings). Participants will be contacted via email each day (at approximately 6 am) to invite them to complete the survey for that day of the study protocol.

For subsequent days (days 1-6, 8-13, 15-20) participants will be contacted and asked to complete a daily survey which will assess their previous day use of LCCs, as well as cigarettes and e-cigarettes. During these daily surveys, participants assigned to condition 1 or 2 (i.e., the warning conditions) will view an image of a little cigar and cigarillo package with a warning according to the participant's condition. Participants within each warning condition will view a total of 6 different warnings over the course of 6 days each week, this will be repeated 3 times during the study, resulting in a total of 18 exposures. Participants will be required to view the warning for at least 5 seconds before answering questions.

On days 7 and 14 participants will be asked to complete a slightly longer survey with questions about their LCC behaviors including the number of LCCs used in the past week, the number of LCCs butted out because they wanted to smoke less, the number of LCCs forgone, other tobacco use, blunt use, and quit intentions and attempts.

For the post-test on day 21, participants will be asked to complete a longer questionnaire about their current tobacco use and behaviors including current LCC smoking behavior, LCC nicotine dependence, other tobacco product (OTP) use, LCC and OTP quit intentions, and LCC and O

ELIGIBILITY:
Inclusion Criteria:

* Members of the recruitment panel (the investigators are partnering with a panel provider for recruitment of all participants)
* Agree to provide their honest answers
* Current little cigar and/or cigarillo every day or some day users
* Over 21 years old
* Currently living in US
* Feel comfortable taking a survey in English without help
* Feel comfortable taking an online survey without help
* Have an email address that they check regularly
* Have access to the internet at work or home
* Able to read and respond to surveys delivered to their email
* Able to complete 2 surveys that take approximately 20 minutes
* Able to complete a 5 minute survey each day for 20 days
* Able to verify they are not a bot using CAPTCHA
* Able to answer a simple, random math question

Exclusion Criteria:

* None

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1029 (Actual)
Dates: Start 2023-05-22 (Actual); Primary Completion 2023-08-27 (Actual); Study Completion 2023-08-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adam O Goldstein, Principal Investigator — the University of North Carolina (UNC) Department of Family Medicine
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make data collection instruments available for public use after data collection and analyses are complete. On request, the investigators will also make data sets available, stripped of individual identifiers, following publication of the study's main findings.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The supporting documents and data will become available when study results are submitted to ClinicalTrials.gov. Deidentified study data sets will be available, by request, following publication of the study's main findings.
Access Criteria: The investigators will decide whether to share deidentified study data sets on a case by case basis, and will prioritize sharing the data sets with qualified tobacco regulatory science researchers.

REFERENCES:
- [Derived] Goldstein AO, Jarman KL, Ranney LM, Cornacchione Ross J, Kowitt SD, Enyioha C, Clark SA, Sheeran P, Thrasher JF, Jenson D, Vielot NA. Little Cigar and Cigarillo Graphic Health Warnings and Quitting Behaviors: A Randomized Clinical Trial. JAMA Netw Open. 2025 Aug 1;8(8):e2526799. doi: 10.1001/jamanetworkopen.2025.26799. PMID 40815515
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited and screened for study eligiblity online between May and August 2024, and invited to in the study once they were determined to be eligible.
Pre-assignment Details: 1,114 potential participants began the baseline survey. Of those, 44 did not consent to participate in the study, and 41 did not complete the baseline questionnaire and were not randomized. 1,029 participants were enrolled and randomized in the study.
Period: Overall Study
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Started | 339 | 346 | 344
Completed | 339 | 346 | 344
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Everyone who enrolled in the study, consented to participate, completed the baseline questionnaire, and was randomized to each condition.
Groups:
- Total: Total of all reporting groups
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention | Total
Number analyzed (Participants) | 339 | 346 | 344 | 1029
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.03 (10.44) | 44.48 (11.73) | 44.07 (11.61) | 43.86 (11.29)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 175 | 208 | 195 | 578
  Female | 163 | 138 | 148 | 449
  Another Gender | 1 | 0 | 1 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 68 | 50 | 52 | 170
  Not Hispanic or Latino | 270 | 294 | 291 | 855
  Unknown or Not Reported | 1 | 2 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 5 | 4 | 1 | 10
  Asian | 21 | 13 | 19 | 53
  Native Hawaiian/Pacific Islander | 0 | 1 | 1 | 2
  Black/African American | 70 | 70 | 77 | 217
  White | 203 | 228 | 214 | 645
  More than one Race | 24 | 20 | 21 | 65
  Unknown not reported | 16 | 10 | 11 | 37
Region of Enrollment [Number; unit: participants]
  United States | 339 | 346 | 344 | 1029

OUTCOME MEASURES:

1. Primary Outcome: LCC Quit Intentions
Description: Average quit intention score measured by survey. Quit intention measured with 3 questions, the final quit intention score is a mean of the response to the 3 questions, on a scale of 1 to 4, where 1 indicates low intention to quit, and 4 indicates a high intention to quit.
Time Frame: day 21 (post test)
Population: Participants who responded to the scale at the time point of interest, post test on day 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 311 | 317 | 312
score on a scale | 2.9 (1.10) | 2.49 (1.12) | 2.54 (1.09)

2. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant.
Time Frame: day 1
Population: Participants who responded to the measures at the time point of interest, day 1
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 264 | 268 | 255
number of LCCs | 2.75 (4.09) | 2.47 (3.14) | 2.28 (2.85)

3. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 2
Population: Participants who responded to the measures at the time point of interest, day 2
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 268 | 271 | 278
number of LCCs | 2.43 (3.09) | 2.62 (3.30) | 2.21 (2.79)

4. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day was reported by participants.
Time Frame: day 3
Population: Participants who responded to the measures at the time point of interest, day 3
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 279 | 258 | 264
number of LCCs | 2.56 (3.17) | 2.66 (3.13) | 2.44 (2.86)

5. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant.
Time Frame: day 4
Population: Participants who responded to the measures at the time point of interest, day 4
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 275 | 294 | 289
number of LCCs | 2.66 (3.51) | 3.04 (4.46) | 2.50 (2.95)

6. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 5
Population: Participants who responded to the measures at the time point of interest, day 5
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 283 | 282 | 273
number of LCCs | 2.77 (3.67) | 3.07 (4.21) | 2.43 (2.78)

7. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 6
Population: Participants who responded to the measures at the time point of interest, day 6
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 295 | 301 | 291
number of LCCs | 2.66 (3.72) | 3.12 (4.81) | 2.20 (2.64)

8. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 298 | 299 | 293
number of LCCs | 2.30 (3.18) | 2.73 (4.04) | 2.33 (3.49)

9. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 8
Population: Participants who responded to the measures at the time point of interest, day 8
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 294 | 299 | 294
number of LCCs | 2.37 (3.61) | 2.68 (4.46) | 2.28 (3.13)

10. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 9
Population: Participants who responded to the measures at the time point of interest, day 9
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 293 | 292 | 298
number of LCCs | 2.64 (4.28) | 2.68 (4.50) | 2.43 (3.27)

11. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 10
Population: Participants who responded to the measures at the time point of interest, day 10
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 284 | 298 | 284
number of LCCs | 2.62 (4.50) | 2.56 (4.16) | 2.39 (3.27)

12. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 11
Population: Participants who responded to the measures at the time point of interest, day 11
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 280 | 288 | 284
number of LCCs | 2.69 (4.11) | 2.94 (4.47) | 2.47 (3.23)

13. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 12
Population: Participants who responded to the measures at the time point of interest, day 12
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 285 | 293 | 284
number of LCCs | 2.28 (3.28) | 2.77 (4.33) | 2.46 (3.01)

14. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 13
Population: Participants who responded to the measures at the time point of interest, day 13
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 291 | 297 | 295
number of LCCs | 2.62 (3.86) | 2.79 (4.61) | 2.50 (3.38)

15. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 278 | 293 | 288
number of LCCs | 2.19 (3.24) | 2.44 (4.58) | 2.24 (3.47)

16. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 15
Population: Participants who responded to the measures at the time point of interest, day 15
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 268 | 274 | 267
number of LCCs | 2.35 (4.27) | 2.56 (4.46) | 2.26 (3.39)

17. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 16
Population: Participants who responded to the measures at the time point of interest, day 16
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 274 | 290 | 283
number of LCCs | 2.21 (3.07) | 2.62 (4.43) | 2.35 (3.57)

18. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 17
Population: Participants who responded to the measures at the time point of interest, day 17
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 279 | 290 | 286
number of LCCs | 2.23 (3.38) | 2.62 (4.35) | 2.38 (3.58)

19. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 18
Population: Participants who responded to the measures at the time point of interest, day 18
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 279 | 277 | 272
number of LCCs | 2.26 (3.33) | 2.87 (4.51) | 2.47 (3.36)

20. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 19
Population: Participants who responded to the measures at the time point of interest, day 19
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 273 | 289 | 284
number of LCCs | 2.27 (3.38) | 2.85 (4.36) | 2.38 (3.39)

21. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 20
Population: Participants who responded to the measures at the time point of interest, day 20
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 288 | 289 | 283
number of LCCs | 2.18 (3.46) | 2.62 (4.25) | 2.36 (3.40)

22. Secondary Outcome: Number of LCCs Smoked in Past Day
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past day reported by participant
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 305 | 311 | 306
number of LCCs | 2.13 (3.30) | 2.34 (3.36) | 2.43 (4.58)

23. Secondary Outcome: Number of Days Smoked LCCs in Past Week
Description: The mean number days that a participant reported smoking little cigars and cigarillos (LCCs) smoked in the past week
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 307 | 305 | 302
number of days | 3.46 (2.29) | 3.58 (2.31) | 3.46 (2.25)

24. Secondary Outcome: Number of Days Smoked LCCs in Past Week
Description: The mean number days that a participant reported smoking little cigars and cigarillos (LCCs) smoked in the past week
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 286 | 300 | 295
number of days | 3.26 (2.40) | 3.50 (2.38) | 3.45 (2.28)

25. Secondary Outcome: Number of Days Smoked LCCs in Past Week
Description: The mean number days that a participant reported smoking little cigars and cigarillos (LCCs) smoked in the past week
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: number of days
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 312 | 317 | 313
number of days | 3.15 (2.44) | 3.46 (2.47) | 3.41 (2.29)

26. Secondary Outcome: Number of LCCs Smoked in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past week reported by participant
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 307 | 305 | 302
number of LCCs | 15.66 (23.13) | 16.05 (24.84) | 13.32 (17.32)

27. Secondary Outcome: Number of LCCs Smoked in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past week reported by participant
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 286 | 300 | 295
number of LCCs | 14.67 (22.45) | 15.35 (22.37) | 13.47 (18.03)

28. Secondary Outcome: Number of LCCs Smoked in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) smoked in the past week reported by participant
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 311 | 317 | 313
number of LCCs | 14.11 (20.30) | 15.89 (22.38) | 13.93 (18.94)

29. Secondary Outcome: Number of LCCs Butted Out in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported butting out in the past week
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 300 | 298 | 293
number of LCCs | 4.24 (7.86) | 3.64 (18.09) | 3.03 (6.51)

30. Secondary Outcome: Number of LCCs Butted Out in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported butting out in the past week
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 276 | 295 | 287
number of LCCs | 3.11 (5.22) | 3.48 (15.53) | 2.59 (5.71)

31. Secondary Outcome: Number of LCCs Butted Out in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported butting out in the past week
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 304 | 311 | 305
number of LCCs | 3.11 (5.41) | 3.46 (14.93) | 2.81 (5.67)

32. Secondary Outcome: Number of LCCs Forgone in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported forgoing in the past week
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 307 | 305 | 302
number of LCCs | 3.85 (5.24) | 3.64 (17.62) | 2.88 (4.83)

33. Secondary Outcome: Number of LCCs Forgone in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported forgoing in the past week
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 286 | 300 | 295
number of LCCs | 6.79 (30.85) | 3.47 (15.39) | 2.81 (4.31)

34. Secondary Outcome: Number of LCCs Forgone in the Past Week
Description: The mean number of little cigars and cigarillos (LCCs) that participants reported forgoing in the past week
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: number of LCCs
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 311 | 317 | 313
number of LCCs | 5.69 (14.67) | 4.30 (15.95) | 3.46 (7.30)

35. Secondary Outcome: LCC Quit Attempts in Past Week
Description: The number and percent of participants who reported trying to quit smoking little cigars and cigarillos (LCCs) in the past week
Time Frame: day 7
Population: Participants who responded to the measures at the time point of interest, day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 307 | 305 | 301
Participants | 108 | 61 | 62

36. Secondary Outcome: LCC Quit Attempts in Past Week
Description: as for outcome 35
Time Frame: day 14
Population: Participants who responded to the measures at the time point of interest, day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 286 | 299 | 295
Participants | 102 | 71 | 66

37. Secondary Outcome: LCC Quit Attempts in Past Week
Description: as for outcome 35
Time Frame: day 21 (post test)
Population: Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Count of Participants; unit: Participants
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 311 | 317 | 312
Participants | 134 | 90 | 86

38. Secondary Outcome: LCC Quit Intentions
Description: as for outcome 1
Time Frame: day 7
Population: Participants who responded to the scale at the time point of interest, day 7
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 307 | 305 | 301
score on a scale | 2.76 (1.07) | 2.33 (1.05) | 2.46 (1.04)

39. Secondary Outcome: LCC Quit Intentions
Description: as for outcome 1
Time Frame: day 14
Population: Participants who responded to the scale at the time point of interest, day 14
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
Number analyzed (Participants) | 286 | 299 | 295
score on a scale | 2.82 (1.08) | 2.42 (1.09) | 2.51 (1.04)

40. Secondary Outcome: Self Reported Learning
Description: Mean self-reported learning reported by participants. Self-reported learning measured with one item on a 1 to 5 scale, where 1 indicates no learning, and 5 indicates a great deal of learning from the warnings in the study. Self reported learning is only measured in conditions 1 and 2, the conditions that receive warnings.
Time Frame: day 21 (post test)
Population: Only Newly developed warnings with images and FDA proposed text-only warnings were included. Participants who responded to the measures at the time point of interest, day 21 (post test)
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings
Number analyzed (Participants) | 311 | 316
units on a scale | 4.14 (1.01) | 3.60 (1.18)

ADVERSE EVENTS:
Time Frame: Low risk study, no adverse event data collected
Description: Low risk study, no adverse event data collected
Arm/Group | Newly Developed Warnings With Images | FDA Proposed Text-only Warnings | Control Group, no Intervention
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-04-17): https://cdn.clinicaltrials.gov/large-docs/51/NCT05849051/Prot_SAP_ICF_000.pdf